CLINICAL TRIAL: NCT07020936
Title: Safety and Feasibility Testing of AIDANET in Children Age 6-13 Years
Brief Title: AIDANET Pediatrics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mark D. DeBoer, MD, MSc., MCR (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mark D. DeBoer, MD, MSc., MCR, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 302210
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Adaptive NETwork (AIDANET) system; Fully Closed Loop (FCL); Specifically modified Mobi system
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This study is a randomized crossover, device safety/feasibility trial with a supervised house/hotel with transition to home use, interventional trial of AIDANET.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Usual Care before experimental system; system with Normal Glycemia Goal (Other): Participants will complete two weeks Usual Care Control Period before the use of the AIDANET system, with system employing Normal Glycemia Goal.
  Interventions: Device: Normal Glycemia Goal
- Usual Care before experimental system; system with Tight Glycemia Goal (Other): Participants will complete two weeks Usual Care Control Period before the use of the AIDANET system, with system employing Tight Glycemia Goal.
  Interventions: Device: Tight Glycemia Goal
- Usual Care after experimental system; system with Normal Glycemia Goal (Other): Participants will complete two weeks Usual Care Control Period after the use of the AIDANET system, with system employing Normal Glycemia Goal.
  Interventions: Device: Normal Glycemia Goal
- Usual Care after experimental system; system with Tight Glycemia Goal (Other): Participants will complete two weeks Usual Care Control Period after the use of the AIDANET system, with system employing Tight Glycemia Goal.
  Interventions: Device: Tight Glycemia Goal

INTERVENTIONS:
Device: Normal Glycemia Goal — Participants will use the normal AIDANET system aggressivity adjustment to achieve target glucose for both the hotel and AIDANET at home periods.
  Arms: Usual Care after experimental system; system with Normal Glycemia Goal; Usual Care before experimental system; system with Normal Glycemia Goal
Device: Tight Glycemia Goal — Participants will have the AIDANET system controller target set to have higher aggressivity adjustment to maintain target glucose for both the hotel and AIDANET at home periods.
  Arms: Usual Care after experimental system; system with Tight Glycemia Goal; Usual Care before experimental system; system with Tight Glycemia Goal

SUMMARY:
AIDANET algorithm with smart-phone based control system (study smart phone), specifically modified Tandem insulin system (study insulin pump), and Dexcom G6 CGM (study CGM).

DETAILED DESCRIPTION:
This study aims to demonstrate the safety and feasibility of the Automated insulin delivery as Adaptive NETwork (AIDANET) system among children age 6-13 years. This includes use of new features allowing requested correction boluses and setting a tighter glycemia goal.

The proposed work is a safety and feasibility study of the FCL system and is not intended to be powered to fully demonstrate efficacy of the system. The sample size of up to 24 completed participants was selected based on previous experience of the feasible number of individuals to supervise at one time under similar study conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥6.0 and ≤13 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
3. Currently using insulin pump for at least three months; Any pump, either open loop or hybrid closed loop may be used.
4. Currently using insulin for at least six months.
5. Willingness to use lispro/aspart in the insulin pump during the study.
6. Currently using a Dexcom G6 or G7 CGM.
7. Has one or more parent/guardian knowledgeable about emergency procedures for severe hypoglycemia and able to contact emergency services and study staff that live with participant.
8. Participant not currently known to be pregnant or breastfeeding.
9. If participant capable of becoming pregnant, must agree to use a form of contraception to prevent pregnancy while a participant in the study (e.g. hormonal contraception, abstinence from heterosexual intercourse). A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
10. Willingness to use the study FCL system (CGM, pump, and phone) during the relevant study period.
11. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.
12. Willingness to participate in all study procedures including the house/hotel session and to consume approximately 3 unannounced meals per day during the relevant portion of the supervised hotel session.
13. Access to internet at-home and willingness to upload data during the study as needed.
14. Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol.
15. Participant is proficient in reading and writing English.

Exclusion Criteria:

1. Plans to start a new non-insulin glucose-lowering agent (e.g., GLP-1 receptor agonists, Symlin, DPP-4 inhibitors, sulfonylureas). Participants may be on a stable dose of such an agent for at least the past month.
2. Current use of an SGLT-2 or SGLT-1/2 inhibitor due to risk of euglycemic Diabetic ketoacidosis (DKA).
3. Hemophilia or any other bleeding disorder.
4. History of severe hypoglycemic events with seizure or loss of consciousness in the last 6 months.
5. History of diabetic ketoacidosis (DKA) event in the last 6 months.
6. History of chronic renal disease (Stage 4 or unstable Stage 3b per investigator judgment) or currently on peritoneal or hemodialysis.
7. History of adrenal insufficiency.
8. Currently being treated for a seizure disorder.
9. Hypothyroidism or hyperthyroidism that is not adequately treated.
10. Coronary artery disease or other heart condition that would prevent participation in moderate intensity exercise.
11. Use of oral or injectable steroids at the time of enrollment or within the last 4 weeks.
12. Planned surgery during the study period.
13. Known ongoing adhesive intolerance that is not well managed.
14. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk.
15. Participation in another interventional trial at the time of enrollment.
16. Participant with a direct supervisor involved in the conduct of the trial.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of mean CGM between FCL and Usual Care | 28 days
  Non-inferiority of the mean CGM between the two weeks of the Usual Care observational period and the two weeks of AIDANET at-home

SECONDARY OUTCOMES:
GMI derived from mean CGM | 28 days
  Non-inferiority of GMI derived from the mean CGM between the two weeks of the Usual Care observational period and the two weeks of AIDANET at-home
Time in range 70-180 mg/dL | 28 days
  Non-inferiority of time in range 70-180 mg/dL between the two weeks of the Usual Care observational period and the two weeks of AIDANET at-home
CGM standard deviation (StDev) | 28
  Non-inferiority of CGM standard deviation (StDev) between the two weeks of the Usual Care observational period and the two weeks of AIDANET at-home
CGM coefficient of variation (CV) | 28 days
  Non-inferiority of CGM coefficient of variation (CV) between the two weeks of the Usual Care observational period and the two weeks of AIDANET at-home
CGM %<54 mg/dL | 28 days
  Non-inferiority of CGM %<54 mg/dL between the two weeks of the Usual Care observational period and the two weeks of AIDANET at-home
CGM %<70 mg/dL | 28 days
  Non-inferiority of CGM %<70 mg/dL between the two weeks of the Usual Care observational period and the two weeks of AIDANET at-home
CGM %>180 mg/dL | 28 days
  Non-inferiority of CGM %>180 mg/dL between the two weeks of the Usual Care observational period and the two weeks of AIDANET at-home
CGM %>250 mg/dL | 28 days
  Non-inferiority of CGM %>250 mg/dL between the two weeks of the Usual Care observational period and the two weeks of AIDANET at-home
Non-inferiority of mean CGM between Normal Glycemia Goal and Tight Glycemia Goal | 17 days
  Mean CGM and other outcomes listed above will be assessed between Normal Glycemia Goal and Tight Glycemia Goal groups

CONTACTS AND LOCATIONS:
Overall Officials: Mark DeBoer, MD, Study Chair — University of Virginia Center for Diabetes Technology
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available after publication of the primary publications of the study
Access Criteria: The data sharing agreements will be formulated by the study team.